CLINICAL TRIAL: NCT04829201
Title: Virtual Surgery of the Upper Airways-New Solutions to Obstructive Sleep Apnea Treatment
Brief Title: Virtual Surgery of the Upper Airways
Acronym: VirtuOSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: SINTEF Health Research (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RCN303218
Record Dates: First submitted 2021-02-08; First posted 2021-04-02 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Surgery; Rhinoplasty; Nasal Obstruction; Soft tissue biomechanics
MeSH Terms: conditions — Sleep Apnea, Obstructive; Nasal Obstruction | interventions — Orthognathic Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Soft tissue specimen from upper airways; soft palate and tonsils
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obstructive sleep apnea (OSA): OSA patients who are eligible for either functional septorhinoplasty or oropharyngeal/orthognathic surgery
  Interventions: Procedure: functional septorhinoplasty or oropharyngeal/orthognathic surgery

INTERVENTIONS:
Procedure: functional septorhinoplasty or oropharyngeal/orthognathic surgery — obtain pre- and postoperative data in order to describe the specific changes in airflow and upper soft tissue behavior that causes sleep apnea

SUMMARY:
Obstructive sleep apnea (OSA) is a sleep related breathing disorder caused by repetitive collapses of the upper airways resulting in impaired breathing, oxygen desaturation and sleep disturbances. OSA has a massive impact on global health contributing directly to cardiovascular diseases, insulin resistance, metabolic syndrome and daytime fatigue and is repeatedly associated with an increase in motor vehicle accidents.

The mainstay of treatment is still the use of positive airway pressure or surgery of the upper airways, but the success rate is persistently low. Surgery may be of help, but there is a lack of patient-specific options in both diagnostics and treatment.

Mathematical and computational modeling is expected to provide significant insight into the airway function and onset of OSA.

This study is part of a project that will rely on biomedical engineering to obtain the required insight to produce software tools for computer-aided diagnostics and treatment of OSA.

DETAILED DESCRIPTION:
This study is the clinical part of a project that contains 4 work packages (WP 1-4). The clinical study (work WP 1) will ensure the inclusion of up to 30 patients with verified sleep apnea that will be in need of either structural nasal surgery, pharyngeal surgery or orthognathic surgery. Studies of nasal airflow and pressure as well as a detailed ConeBeam CT scans of the upper airways will be performed before and after surgery.

WP 2, 3 and 4 deals with the mathematical modeling, structural mechanic modeling and the patient-specific airflow modeling.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnea
* need either functional septorhinoplasty or oropharyngeal/orthognathic surgery in order to establish adequate airway patency
* have undergone sleep registration using polysomnography and ultrawideband radar
* on the subsequent clinical evaluation presenting either 1) intranasal obstruction, due to malalignment of the nasal septal cartilage or the nasal outer framework; and/or 2) oropharyngeal obstruction or retrognathia.

Exclusion Criteria:

* previous nasal or oropharyngeal surgery
* previous use of nasal decongestant or nasal topical steroids over the last 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients within the community of Mid-Norway referred to the sleep clinic from primary or secondary care facilities.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Apnea-Hypopnea Index (AHI) | Baseline and 3 months postoperatively
  AHI is measured by sleep polygraphy in all patients before and after surgery
Upper airway soft tissue characteristics | Up to 3 months postoperatively
  Specific descriptions of deformation and strain in soft tissues in sleep apnea patients

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn H Skallerud, phd prof, Study Director — NTNU, Fac IV, Dept of Structural Engineering; Ståle Nordgård, phd prof, Principal Investigator — NTNU, Fac MH, Dept of Neuromedicine and Movement Science; Bernhard Müller, phd prof, Principal Investigator — NTNU, Fac IV, Dept of Energy and Process Engineering; Sverre G Johnsen, phd, Principal Investigator — SINTEF Health Research; Ståle Nordgård, phd prof, Study Director — St Olavs Hospital, Clinic Ear Nose and Throat
Locations (2):
- Norway (2):
  - St Olavs Hospital, Trondheim, Trøndelag
  - Aleris Solsiden, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: third quarter 2022 until the end of 2024
Access Criteria: links to all publications will be made available on the website
URL: http://osas.no